CLINICAL TRIAL: NCT00929617
Title: Enhancing Physical Activity Adherence After Breast Cancer Diagnosis (BEAT Cancer Study II)
Brief Title: Enhancing Physical Activity Adherence After Breast Cancer Diagnosis (BEAT Cancer II)
Acronym: BEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); University of Illinois at Urbana-Champaign (Other); Southern Illinois University (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROG-SCCI 09-003-2; 3R01CA136859-02S1 (NIH); U01CA136859 (NIH)
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; physical activity; exercise; quality of life; doubly labeled water
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: exercise with 2 counseling types (Experimental): Patients will participate in 12 individual exercise sessions with an exercise specialist; plus attend 6 discussion group sessions with a trained facilitator; plus 3 face-to-face, individual counseling sessions with an exercise specialist
  Interventions: Behavioral: Experimental 1: exercise with 2 counseling types
- 2. Usual Care - written materials (Other): Patients will receive written materials about exercise for cancer survivors
  Interventions: Other: Usual Care - written materials

INTERVENTIONS:
Behavioral: Experimental 1: exercise with 2 counseling types — Patients will participate in 12 individual exercise sessions with an exercise specialist which will include stretching exercises and aerobic treadmill walking; plus attend 6 discussion group sessions with a trained facilitator; plus 3 face-to-face, individual counseling sessions with an exercise specialist
  Arms: 1: exercise with 2 counseling types
Other: Usual Care - written materials — Patients will receive written materials about exercise for cancer survivors
  Arms: 2. Usual Care - written materials

SUMMARY:
The purpose of the study is to compare the effects of one exercise/counseling protocol with usual care on long term exercise adherence and on changes in health related outcomes after breast cancer diagnosis.

DETAILED DESCRIPTION:
Physical activity may improve quality of life, the control of comorbid conditions, and weight management while reducing breast cancer recurrence and mortality among breast cancer survivors. Unfortunately, most breast cancer survivors do not engage in regular physical activity. In fact, breast cancer survivors are often less active after a diagnosis and may not return to pre-diagnosis activity levels. Therefore, we conducted a pilot study, "BEAT Cancer", to test a specifically defined physical activity behavior change intervention to increase physical activity for breast cancer survivors. The pilot study showed significant improvement in both physical activity and health outcomes for the study participants after the intervention. Importantly, the pilot intervention resulted in changes in physical activity and social cognitive theory constructs, such as the participants feeling more confident in their ability to exercise. The positive results enhance our potential for testing mechanisms that encourage physical activity behavior change in breast cancer survivors. The current study is a follow-up to confirm program effectiveness at 3 months and to test sustainability of results at 3-12 months. We propose a multi-center, randomized controlled trial enrolling 356 breast cancer survivors with the following study aims:

1. To compare the effects of the 3-month BEAT Cancer physical activity behavior change intervention to usual care on short and longer term physical activity adherence among breast cancer survivors. We hypothesize that, compared with usual care, the intervention will result in a significant increase in physical activity after the intervention that will be maintained up to 12 months after baseline.
2. To better understand the reasons why breast cancer patients change their physical activity behavior, we will compare the effects of the BEAT Cancer physical activity behavior change intervention to usual care on social cognitive factors to see if such changes contribute to physical activity behavior change. We hypothesize that, compared with usual care, the intervention will result in significant improvements in social cognitive factors which lead to changes in physical activity behavior.
3. We also aim to compare the short and longer term health effects of the BEAT Cancer physical activity behavior change intervention when compared with usual care. We hypothesize that, compared with usual care, the intervention will result in significant improvements in fitness, muscle strength, waist-to-hip ratio, quality of life, fatigue, and sleep quality, while reducing joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients between the ages of 18 and 70 years of age with a diagnosis of ductal carcinoma in situ (DCIS) or Stage I, II, or IIIA breast cancer and who are not currently receiving (and do not plan to receive during the duration of the study) chemotherapy or radiation therapy. The participant may be taking longer term therapies such as aromatase inhibitors, estrogen receptor modulators, etc. The upper age limit of 70 years was chosen to reduce the likelihood of adverse events or study drop-out due to increasing comorbidities (e.g., cardiovascular disease) that occur with age.
* If the patient has undergone a surgical procedure, enrollment will be delayed until ≥ 8 weeks post-procedure.
* English speaking.
* Medical clearance for participation provided by primary care physician or oncologist.
* Participating, on average, in no more than 60 minutes of moderate physical activity or no more than 30 minutes of vigorous activity per week during the past six months.

Exclusion Criteria:

* Diagnosis of dementia or organic brain syndrome.
* Medical, psychological, or social characteristic that would interfere with ability to fully participate in program activities and assessments (e.g., psychosis, schizophrenia, etc.).
* Contraindication to participation in a regular physical activity program.
* Metastatic or recurrent disease.
* Inability to ambulate.
* Anticipates undergoing elective surgery during the duration of the intervention which would interfere with intervention participation (e.g., breast reconstructive surgery).
* Planned travel that would interfere with scheduled study sessions (no travel in the 1st 4 months and no travel ≥ 1 week in the last 8 weeks of the intervention).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2009-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
change in physical activity | baseline to 3 months
  Physical activity will be measured with accelerometers and self-report questionnaire. Change will be calculated as difference between baseline and 3 endpoints (3, 6 and 12 months).
change in physical activity | 3 mos to 6 months
  Physical activity will be measured with accelerometers and self-report questionnaire. Change will be calculated as difference between baseline and 3 endpoints (3, 6 and 12 months).
change in physical activity | 6 months to 12 months
  Physical activity will be measured with accelerometers and self-report questionnaire. Change will be calculated as difference between baseline and 3 endpoints (3, 6 and 12 months).

SECONDARY OUTCOMES:
change in treadmill fitness | baseline, 3 months, 6 months, 12 months
  Treadmill fitness will be measured by sub-maximal fitness test. Change will be calculated as difference between baseline and 3 endpoints (3, 6 and 12 months).
change in waist-to-hip ratio | baseline, 3 months, 6 months, 12 months
  Waist-to-hip ratio will be measured with a tape measure. Change will be calculated as difference between baseline and 3 endpoints (3, 6 and 12 months).
change in 3-day dietary intake | baseline, 3 months, 6 months, 12 months
  3-day dietary intake will be measured by questionnaire. Change will be calculated as difference between baseline and 3 endpoints (3, 6 and 12 months).

OTHER OUTCOMES:
Energy expenditure (doubly labeled water) | baseline, 3 months, and 6 months
  Doubly labeled water results will be used to determine reliability of accelerometer measures as part of an NCI funded supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q. Rogers, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Illinois, Champaign, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois

REFERENCES:
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Markwell S, Pamenter R, Courneya KS, Hoelzer K, Naritoku C, Edson B, Jones L, Dunnington G, Verhulst S. Physical activity and health outcomes three months after completing a physical activity behavior change intervention: persistent and delayed effects. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1410-8. doi: 10.1158/1055-9965.EPI-08-1045. Epub 2009 Apr 21. PMID 19383889
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Pamenter R, Courneya KS, Markwell S, Verhulst S, Hoelzer K, Naritoku C, Jones L, Dunnington G, Lanzotti V, Wynstra J, Shah L, Edson B, Graff A, Lowy M. A randomized trial to increase physical activity in breast cancer survivors. Med Sci Sports Exerc. 2009 Apr;41(4):935-46. doi: 10.1249/MSS.0b013e31818e0e1b. PMID 19276838
- [Background] Rogers LQ, Markwell SJ, Verhulst S, McAuley E, Courneya KS. Rural breast cancer survivors: exercise preferences and their determinants. Psychooncology. 2009 Apr;18(4):412-21. doi: 10.1002/pon.1497. PMID 19241491
- [Background] Rogers LQ, Courneya KS, Verhulst S, Markwell SJ, McAuley E. Factors associated with exercise counseling and program preferences among breast cancer survivors. J Phys Act Health. 2008 Sep;5(5):688-705. doi: 10.1123/jpah.5.5.688. PMID 18820344
- [Background] Rogers LQ, McAuley E, Courneya KS, Verhulst SJ. Correlates of physical activity self-efficacy among breast cancer survivors. Am J Health Behav. 2008 Nov-Dec;32(6):594-603. doi: 10.5555/ajhb.2008.32.6.594. PMID 18442339
- [Background] Rogers LQ, Markwell S, Hopkins-Price P, Vicari S, Courneya KS, Hoelzer K, Verhulst S. Reduced barriers mediated physical activity maintenance among breast cancer survivors. J Sport Exerc Psychol. 2011 Apr;33(2):235-54. doi: 10.1123/jsep.33.2.235. PMID 21558582
- [Background] Rogers LQ, McAuley E, Anton PM, Courneya KS, Vicari S, Hopkins-Price P, Verhulst S, Mocharnuk R, Hoelzer K. Better exercise adherence after treatment for cancer (BEAT Cancer) study: rationale, design, and methods. Contemp Clin Trials. 2012 Jan;33(1):124-37. doi: 10.1016/j.cct.2011.09.004. Epub 2011 Sep 29. PMID 21983625
- [Result] Rogers LQ, Courneya KS, Anton PM, Hopkins-Price P, Verhulst S, Vicari SK, Robbs RS, Mocharnuk R, McAuley E. Effects of the BEAT Cancer physical activity behavior change intervention on physical activity, aerobic fitness, and quality of life in breast cancer survivors: a multicenter randomized controlled trial. Breast Cancer Res Treat. 2015 Jan;149(1):109-19. doi: 10.1007/s10549-014-3216-z. Epub 2014 Nov 23. PMID 25417174
- [Derived] Rogers LQ, Midthune D, Dodd K, Bowles H, McAuley E, Courneya KS, Barrett B, Razis S, Hunter GR, Carter SJ, Carroll RJ, Kipnis V. Accelerometer measurement error in a randomized physical activity intervention trial in breast cancer survivors was nondifferential but attenuated the intervention effect. Int J Behav Nutr Phys Act. 2025 May 26;22(1):59. doi: 10.1186/s12966-025-01760-5. PMID 40420153
- [Derived] Schleicher E, McAuley E, Courneya KS, Anton P, Ehlers DK, Phillips SM, Brown NI, Oster RA, Pekmezi D, Rogers LQ. Breast cancer survivors' exercise preferences change during an exercise intervention are associated with post-intervention physical activity. J Cancer Surviv. 2024 Oct;18(5):1453-1463. doi: 10.1007/s11764-023-01389-y. Epub 2023 Apr 29. PMID 37120460
- [Derived] Rogers LQ, Courneya KS, Oster RA, Anton PM, Phillips S, Ehlers DK, McAuley E. Physical activity intervention benefits persist months post-intervention: randomized trial in breast cancer survivors. J Cancer Surviv. 2023 Dec;17(6):1834-1846. doi: 10.1007/s11764-022-01329-2. Epub 2023 Feb 1. PMID 36723801
- [Derived] Schleicher E, McAuley E, Courneya KS, Anton P, Ehlers DK, Phillips SM, Brown NI, Oster RA, Pekmezi D, Rogers LQ. Breast Cancer Survivors' Exercise Preferences Change During an Exercise Intervention and are associated with Post-Intervention Physical Activity. Res Sq [Preprint]. 2023 Jan 20:rs.3.rs-2488848. doi: 10.21203/rs.3.rs-2488848/v1. PMID 36711885
- [Derived] Schleicher E, McAuley E, Courneya KS, Anton P, Ehlers DK, Phillips SM, Oster RA, Pekmezi D, Rogers LQ. Moderators of physical activity and quality of life response to a physical activity intervention for breast cancer survivors. Support Care Cancer. 2022 Dec 17;31(1):53. doi: 10.1007/s00520-022-07477-6. PMID 36526826
- [Derived] Ainsworth MC, Pekmezi D, Bowles H, Ehlers D, McAuley E, Courneya KS, Rogers LQ. Acceptability of a Mobile Phone App for Measuring Time Use in Breast Cancer Survivors (Life in a Day): Mixed-Methods Study. JMIR Cancer. 2018 May 14;4(1):e9. doi: 10.2196/cancer.8951. PMID 29759953
- [Derived] Rogers LQ, Courneya KS, Anton PM, Hopkins-Price P, Verhulst S, Robbs RS, Vicari SK, McAuley E. Social Cognitive Constructs Did Not Mediate the BEAT Cancer Intervention Effects on Objective Physical Activity Behavior Based on Multivariable Path Analysis. Ann Behav Med. 2017 Apr;51(2):321-326. doi: 10.1007/s12160-016-9840-6. PMID 27752993
- See also: National Cancer Institute site on Physical Activity and Cancer — http://www.cancer.gov/cancertopics/factsheet/physical-activity-qa